CLINICAL TRIAL: NCT02822703
Title: Enhancing Relapse Prevention for Smoking Cessation With Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: Enhancing Relapse Prevention for Smoking Cessation With Repetitive Transcranial Magnetic Stimulation
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The City College of New York (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Virginia Tech Carilion School of Medicine and Research Institute (Other)
Responsible Party: Principal Investigator, Christine Sheffer, Associate Medical Professor, The City College of New York
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 639308; R21CA178813 (NIH)
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; tobacco use disorder; delay discounting; repetitive transcranial magnetic stimulation; relapse prevention
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active 20Hz (Experimental): The rTMS device used in this study is the Mastim Super Rapid2 Stimulator with a 70mm Double Air Film Coil. Guidelines indicate that the maximum safe duration of a single train of 20Hz at 110% of the Motor Threshold (MT) is 1.6 seconds. In this study, the stimulator and the coils will be used to stimulate neurons in the left dorsolateral prefrontal cortex (DLPFC), the same location in the brain as that stimulated in the studies supporting the efficacy of this treatment in depression, in order to examine the feasibility of testing this intervention for efficacy in the treatment of tobacco dependence.
  Interventions: Device: rTMS Active 20Hz
- Sham (Sham Comparator): The rTMS sham coil used in this study is manufactured by Magstim and currently classified as an investigational device. There is no intention to treat or prevent a disease and/or alter a function in the body with the sham stimulation provided by the sham coil. In this project, the sham coil will be placed in the same location in the brain as that stimulated in the studies supporting the efficacy of this treatment for depression.
  Interventions: Device: rTMS Sham

INTERVENTIONS:
Device: rTMS Active 20Hz — Active stimulation will be delivered with 70mm Double Air Film Coils. Participants will attend eight 20Hz sessions within two weeks of the scheduled quit date. Participants will receive 20Hz at 110% of the MT for 1 second, less than the limits indicated in the guidelines. These stimulation parameters have been utilized with no serious adverse events in previous studies to decrease delay discounting among smokers and non-smokers. These parameters are similar to or less intense than those utilized in other smoking cessation studies. All participants will receive rTMS over the same area of the DLPFC (6cm anterior to the MT area) while reading relapse prevention booklets supervised by the study coordinator.
  Arms: Active 20Hz
Device: rTMS Sham — The sham stimulation uses a similar 70mm Double Air Film Coil to look and sound like the active coil, but the magnetic field produced by the sham coil is markedly attenuated (only 5% of stimulator output setting: that is 2.25% of the maximum stimulator output (5% of 45% = 2.25%) and biologically inactive. Participants in this condition will attend eight sham sessions within two weeks of their scheduled quit date. During these sessions, they will also read relapse prevention booklets supervised by the study coordinator. The sham coil is not intended to and does not produce a stimulation effect so there is no proposed biologic mechanism of action.
  Arms: Sham

SUMMARY:
Tobacco use is one of the most significant cancer control and public health challenges in the US today. Half of all smokers in the US will attempt to quit tobacco each year, but fully 95% of those who attempt to quit will reverse this decision within 12 months and choose the transient, albeit immediately rewarding activity of smoking at the cost of much larger long-term rewards such as future health and long life. This project seeks to improve scientific knowledge of these decision-making processes and potentially improve the treatment of tobacco dependence by examining the feasibility of using a brain stimulation technique, repetitive Transcranial Magnetic Stimulation or rTMS to improve the efficacy of an existing evidence-based relapse prevention intervention. rTMS is an FDA-cleared treatment for medication resistant depression and is being examined as a treatment for a variety of other disorders. This study will utilize an intensity and duration of rTMS that is well within the safety parameters and similar in location and intensity to that used in previous studies with smokers to reduce cigarette consumption.

DETAILED DESCRIPTION:
This project seeks to improve scientific knowledge of the decision-making processes of smokers and improve tobacco dependence treatments. The dorsolateral prefrontal cortex (DLPFC) influences decision-making by integrating inhibitory mechanisms with emotionally charged information from limbic regions, thereby exerting an inhibitory influence on seductive, immediately rewarding options with long-term costs, such as smoking. Delay discounting is the degree to which one de-values delayed outcomes, such as future health and long life. Converging evidence indicates that choosing a delayed option with a larger reward is associated with increased activity in the DLPFC. This study proposes that choosing to smoke after making a decision to quit reflects a situation where the DLPFC is insufficiently activated to exert an inhibitory influence on the immediately rewarding option of smoking.

Preliminary studies indicate that stimulation of the DLPFC with 20 Hz high frequency repetitive Transcranial Magnetic Stimulation (rTMS) reduces delay discounting (i.e., causes individuals to choose delayed, higher value options); reduces cigarette consumption in smokers intending to quit; improves executive function, learning, memory, and attention; is a promising adjunct to cognitive-behavioral treatment of other disorders; and is likely to improve the efficacy of existing cognitive-behavioral treatments for tobacco dependence.

The goal of this study is to make an informed recommendation, based on measures of feasibility, of whether or not this intervention should be tested for efficacy. A double blind, randomized between-subjects treatment (active or sham) design will be employed in which all subjects are exposed to the same relapse prevention materials during rTMS stimulation.

Aim 1: Examine the feasibility of combining high frequency rTMS with an evidence-based, self-help, cognitive-behavioral relapse prevention intervention using multiple feasibility indicators (demand, acceptability, practicality, limited-efficacy testing, and adequate blinding).

Aim 2: Examine differences in delay discounting between the active and the sham conditions 2, 4, 8, and 12 weeks after the quit day.

Aim 3: Use latency to relapse comparisons to calculate estimates of the effect size of this intervention on abstinence.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old
* Are fluent in English and be able to read English at the 8th grade level
* Pass the Transcranial Magnetic Stimulation Adult Safety and Screening Questionnaire (TASS)
* Report smoking 5-20 cigarettes daily
* Intend to quit smoking in the next 30 days
* Report a motivation level to quit of ≥7 (scale 0-10)
* Pass a urine drug screen for drugs of abuse (marijuana, cocaine, opioids, amphetamines, etc.)
* No plans to move from the area NYC area in the next 4 months and have a consistent, reliable method of communication so that study staff can successfully contact them

Exclusion Criteria:

* self-reported claustrophobia
* personal history of epilepsy
* use of anticonvulsant medication
* head injury, aneurysm, stroke, or previous cranial neurosurgery
* diagnosis of major depressive disorder, bipolar disorder, a schizophrenia-spectrum disorder, tinnitus, or migraines
* metal implants in the head, neck, or cochlea; a pacemaker
* currently taking medications that lower seizure threshold (i.e., such as tricyclic antidepressants or bupropion)
* known pre-existing noise induced hearing loss or concurrent treatment of ototoxic medications (i.e., Aminoglycosides, Cisplatine)
* currently using medications for tobacco cessation (i.e., nicotine replacement, bupropion, varenicline, etc.)
* pregnant or planning to become pregnant in the next 12 weeks
* current regular use of forms of tobacco other than cigarettes

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Latency to relapse | 3.5 months following scheduled quit date
  Abstinence will be assessed with latency to relapse (days from Quit Date to relapse or 7 consecutive days of smoking after a 24 hour quit attempt)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Sheffer, PhD, Principal Investigator — CCNY
Locations (1):
- The City College of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No